CLINICAL TRIAL: NCT05896254
Title: A Phase 1b/2a Randomized, Double-Blind, Placebo-controlled Study of the Safety and Efficacy of MAR001 in Patients With Metabolic Dysfunction
Brief Title: Study of MAR001 in Adults With Metabolic Dysfunction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Marea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAR-102
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MAR001 (Experimental): Subcutaneous injection
  Interventions: Drug: MAR001
- Placebo (Placebo Comparator): Subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MAR001 — Subcutaneous injection
  Arms: MAR001
Drug: Placebo — Subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of multiple doses of MAR001in adult volunteers with metabolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide informed consent and comply with the intervention
* Women of childbearing potential and men agreeing to use an appropriate method of contraception for the duration of the study
* Evidence of metabolic dysfunction at screening (triglyceride levels > 2.8 mmol/L)

Exclusion Criteria:

* Any condition which in the opinion of the investigator prevents the participant from complying with study procedures or prevents the participant from completing the study or interferes with the interpretation of study results
* Pregnant or breastfeeding mothers
* Terminal illness with expected survival of less than 1 year

Note: additional inclusion/exclusion criteria may apply, per protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-07-22 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of MAR001 | 12 weeks
  Incidence and frequency of treatment-emergent adverse events

SECONDARY OUTCOMES:
Effect of MAR001 on triglyceride metabolism | 12 weeks
  Change from baseline in triglyceride levels

CONTACTS AND LOCATIONS:
Overall Officials: Alex DePaoli, Study Director — Marea Tx
Locations (2):
- Australia (2):
  - Brisbane Site, Brisbane
  - Melbourne Site, Melbourne

REFERENCES:
- [Derived] Cummings BB, Joing MP, Bouchard PR, Milton MN, Moesta PF, Ramanan V, Lane A, Hirman J, Trauger JW, Maratos-Flier E, Voznesensky A, Splawski I, Nimonkar AV, Flaherty MM, Yi BA, Meyers D, Huet F, Sahambi SK, Yates DP, Hom D, Hinder M, Basson CT, O'Donnell C, Siegelman ES, Garrett CE, Lehrer-Graiwer J, Juliano RA, Weiss EJ. Safety and efficacy of a novel ANGPTL4 inhibitory antibody for lipid lowering: results from phase 1 and phase 1b/2a clinical studies. Lancet. 2025 May 31;405(10493):1923-1934. doi: 10.1016/S0140-6736(25)00825-6. Epub 2025 May 15. PMID 40383129